CLINICAL TRIAL: NCT00034905
Title: A Comparison of Seroquel vs. Risperidone in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Purpose: Treatment
Other Study IDs: 5077US/0043
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: quetiapine fumarate vs risperidone

SUMMARY:
The purpose of this study is to show equal efficacy of both quetiapine and risperidone in subjects treated with study medication for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria

* Male / Female, 18-65 years old
* Schizophrenia (as per DSM IV)

Exclusion Criteria

* Concurrent use of psychotropic medication
* Does not fulfill moderately ill on CGI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (64):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Anaheim, California
  - Cerritos, California
  - Chula Vista, California
  - Glendale, California
  - Hawthorne, California
  - Long Beach, California
  - San Diego, California
  - Santa Ana, California
  - Torrance, California
  - Farmington, Connecticut
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Miami Beach, Florida
  - North Miami, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Hoffman Estates, Illinois
  - Prairie Village, Kansas
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - New Baltimore, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Reno, Nevada
  - Clementon, New Jersey
  - Lyons, New Jersey
  - Summit, New Jersey
  - Albuquerque, New Mexico
  - Holliswood, New York
  - Montrose, New York
  - New York, New York
  - Oceanside, New York
  - The Bronx, New York
  - White Plains, New York
  - Butner, North Carolina
  - Beachwood, Ohio
  - Chagrin Falls, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Media, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Terrell, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Falls Church, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Kirkland, Washington
  - Tacoma, Washington
  - Vancouver, Washington
  - West Allis, Wisconsin